CLINICAL TRIAL: NCT05661188
Title: Phase II Study of Atezolizumab Plus Tiraglolumab in Combination With Chemoradiotherapy in Localized Squamous Cell Carcinoma of the Anal Canal
Brief Title: Tiraglolumab Atezolizumab and Chemoradiotherapy in Localized Anal Carcinoma (TIRANUS)
Acronym: TIRANUS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Espanol Multidisciplinario del Cancer Digestivo (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEMCAD - 2103 // MO44170
Record Dates: First submitted 2022-11-30; First posted 2022-12-22 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Squamous Cell Carcinoma of the Anal Canal
MeSH Terms: interventions — atezolizumab

STUDY DESIGN:
Intervention Model Description: The TIRANUS trial is a Phase II, single-arm, open-label, non randomized, non controlled, proof-of-concept clinical trial of atezolizumab and tiragolumab in concomitancy with standard chemoradiotherapy (RT, 5-FU, and Cisplatin) as first-line in localized squamous cell carcinoma of the anal canal.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- atezolizumab and tiragolumab in concomitancy with standard chemoradiotherapy (Experimental): TIRANUS is a Phase II, single-arm, open-label, non-randomized, multicenter clinical trial of atezolizumab and tiragolumab in concomitance with standard chemoradiotherapy as first-line in treatment-naïve, localized squamous cell carcinoma of the anal canal who are candidates for radical chemoradiotherapy. Patients with well differentiated stage I anal margin cancer or previously treated with immunotherapy are not eligible.
  All patients receive atezolizumab (1200mg) plus tiragolumab (600 mg) for 2 cycles (Q3W) in concomitance with the 6 weeks of standard scheduled chemoradiotherapy (cisplatin: 60 mg/m² on days 1 and 29; 5-FU: 1000 mg/m² per day on days 1-4 and 29-32; radiotherapy: 1.8 Gy per day / total dose 54 Gy). After the concomitant phase, patients receive atezolizumab and tiragolumab for 6 additional cycles (consolidation phase).
  Interventions: Drug: Atezolizumab plus Tiraglolumab

INTERVENTIONS:
Drug: Atezolizumab plus Tiraglolumab — All patients receive atezolizumab (1200mg) plus tiragolumab (600 mg) for 2 cycles (Q3W) in concomitance with the 6 weeks of standard scheduled chemoradiotherapy (cisplatin: 60 mg/m² on days 1 and 29; 5-FU: 1000 mg/m² per day on days 1-4 and 29-32; radiotherapy: 1.8 Gy per day / total dose 54 Gy). After the concomitant phase, patients receive atezolizumab and tiragolumab for 6 additional cycles (consolidation phase).

SUMMARY:
The peculiarity of anal cancers, with well-established radical chemoradiotherapy that allows tumor-neoantigen formation with platinum-based chemotherapy and radiotherapy with radio-sensitizing chemotherapy could create the perfect environment for immunotherapy in this setting, not only to increase the probability of pathological complete response (CCR) but also creating neoantigen exposure and immune-prevention to reduce the relapse after surgery.

TIRANUS trial is a Phase II, single-arm, open-label, non randomized, non controlled recruiting treatment-naive localized squamous cell carcinoma of the anal canal and are candidates for radical chemoradiotherapy. The trial hypothesizes that the addition of immunotherapy (atezolizumab and tiragolumab) to standard chemoradiotherapy in localized squamous cell carcinoma of the anal canal may improve the CCR at the end of consolidation phase. The study will assess, as the primary endpoint, the CCR, defined as the percentage of patients who have achieved complete response (CR), disappearance of all target lesions and no presence of residual disease assessed by biopsy at the end of consolidation phase. Secondary objectives include survival, safety of the combination, patient reported quality of life, and a substudy of molecular biomarkers determined in tumor biopsy and blood samples.

The main question[s] it aims to answer are:

1. To determine the efficacy of atezolizumab plus tiragolumab concomitantly with chemoradiotherapy in patients with localized squamous cell carcinoma of the anal canal evaluating the clinical response to treatment.
2. To evaluate safety of the intended treatment regimen and Health-related quality of life (HRQoL) in this treatment regimen

All patients will receive atezolizumab plus tiragolumab for 2 cycles in concomitance with the 6 weeks of standard scheduled chemoradiotherapy. (cisplatin, 5-Fluorouracil and radiotherapy). After the concomitant phase, patients will enter a consolidation phase and will receive atezolizumab in combination with tiragolumab up to 24 weeks. Patients will discontinue treatment in case of confirmed progression, toxicity, patient criteria, or physician criteria.

DETAILED DESCRIPTION:
The TIRANUS trial is a Phase II, single-arm, open-label, non randomized, non controlled, proof-of-concept clinical trial of atezolizumab and tiragolumab in concomitancy with standard chemoradiotherapy (RT, 5-Fluorouracil, and Cisplatin) as first-line in localized squamous cell carcinoma of the anal canal.

1. Objectives 1.1 Primary Objectives To determine if atezolizumab plus tiragolumab in concomitancy with chemoradiotherapy is effective in achieving complete remission in patients with localized squamous cell carcinoma of the anal canal assessed by means of clinical complete response (CCR), defined as the percentage of patients who have achieved complete response (CR), disappearance of all lesions according to RECIST 1.1 criteria and no presence of residual disease assessed by biopsy at the end of consolidation phase (week 26).

1.2. Secondary Objectives

Efficacy secondary objectives:

* To evaluate the locoregional failure rate (LFR), defined as the percentage of patients who present progression/relapse of disease in the anal canal and/or regional organs and/or regional lymph nodes. Locoregional failure rate will be estimated using the appropriate logistic regression model at 1-year, 2-years, and 3-years after the first dose of study treatment and end of study.
* To evaluate the disease-free survival (DFS) of patients with localized squamous cell carcinoma of the anal canal, defined as the time elapsed from the first dose of study treatment to progression, relapse, or death from any cause, whichever occurs first. The investigators will assess the DFS rate at 1, 2, and 3 years. The 1-year, 2-years, and 3-years DFS rates are defined as the rate of patients alive and free of relapse or progression at 1, 2, and 3 years after the first dose of study treatment respectively, estimated by Kaplan-Meier.
* To evaluate the colostomy-free survival (CFS) of patients with localized squamous cell carcinoma of the anal canal, defined as the time elapsed from the first dose of study treatment to the date the colostomy was required or death from any cause, whichever occurs first. The 1-year, 2-years, and 3-years CFS rates are defined as the rate of patients alive and free of colostomy at 1, 2, and 3 years after the first dose of study treatment respectively, estimated by Kaplan-Meier.
* To determine the overall survival (OS) of patients with localized squamous cell carcinoma of the anal canal, defined as the time elapsed from the first dose of study treatment until death from any cause. The investigators will assess the OS rate at 3 and 5 years. The 3-years and 5-years OS rates are defined as the rate of patients alive at 3 and 5 years after the first dose of study treatment respectively, estimated by Kaplan-Meier.

Safety secondary objectives

* To evaluate safety of the intended treatment regimen based on the frequency and severity of adverse events and Treatment-emergent adverse events (TEAEs) assessed by NCI CTCAE v5.0.
* Health-related quality of life (HRQoL), assessed through the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C30 (EORTC QLQ-C30) version 3.

Exploratory objectives

* To determine molecular or clinical predictive biomarkers of clinical complete response.
* To evaluate the relationship between the treatment activity and the expression of:

  * Immune checkpoint proteins (including but not limited to PD-1, PD-L1, CD28, OX40, CD40)
  * Presence of infiltrating T cell lymphocytes and immune infiltrate characterization (including but not limited to CD45, CD3, CD8, CD4, CD56, IFNbeta, STAT1, CD 163, H2AX)
  * T-cell clonality (TCR) by multiplex PCR-based clonality (polymerase chain reaction amplification based clonality) // NGS (Next-Generation Sequencing)
  * Tumor mutational burden (TMB) by means of a gene panel with >300 genes.
  * Presence of infections: poliovirus receptor (PVR) and human papillomavirus (HPV)
  * Presence of potential molecular biomarkers in ctDNA (including but not limited to HPV, KRAS, or TP53)

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects ≥ 18 years old.
2. Written informed consent approved by the Independent Ethics Committee (IEC), prior to the performance of any trial activities.
3. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
4. Histologically confirmed squamous cell carcinoma of the anal canal. This may include non-keratinizing histological subtypes (i.e. basaloid, transitional, spheroidal and cloacogenic).
5. Locoregional squamous cell carcinoma of the anal canal with no distant metastasis: stages I, II, IIIA, and IIIB according to the American Joint Cancer Committee (AJCC) Cancer Staging Handbook Seventh Edition (T1-4, N0-1, M0). Patients with well differentiated Stage I anal margin cancer are not eligible.
6. Mandatory archival or recent paraffin-fixed (FFPE) tumor biopsy available at baseline for translational purposes. Fine-needle biopsy is acceptable.

   Note: If there is no archival tumor tissue or not enough tissue available from the biopsy at diagnosis, another biopsy may be requested before treatment begins (after signing the informed consent).
7. At least one evaluable lesion.
8. Patients should meet the criteria for radical chemoradiotherapy for squamous cell carcinoma of the anal canal following international guidelines.
9. Normal life expectancy, excluding cancer mortality risk
10. Patients with adequate normal organ and marrow function assessed within 14 days prior to start of the study treatment as defined below:

    1. Hemoglobin ≥ 9.0 g/dL (Patients may be transfused to meet this criterion).
    2. Absolute neutrophil count (ANC) > 1500 per mm3.
    3. Platelet count ≥ 100,000 per mm3.
    4. Serum total bilirubin ≤ 1.5 X institutional upper limit of normal (ULN). This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of haemolysis or hepatic pathology); however, they will be allowed only in consultation with their physician if total bilirubin ≤ 3 × ULN.
    5. Serum transaminases: alanina aminotransferase (ALT), aspartato aminotransferase (AST) and fosfatase alcalina (ALP) ≤ 2.5X ULN.
    6. Serum albumin ≥ 25 g/L (2.5 g/dL).
    7. Creatinine ≤ 1.5 mg/dL or measured creatinine clearance (CL) > 60 mL/min or Calculated creatinine CL > 60 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for the determination of creatinine clearance:

    Males:

    Creatinine CL (mL/min) = (Weight (kg) × (140 - Age))/ 72 x serum creatinine (mg/dL)

    Females:

    Creatinine CL (mL/min) = ((Weight (kg) × (140 - Age) ×0.85))/72 x serum creatinine (mg/dL)
11. Absence of active infection that requires systemic antibiotics.
12. Female subjects of childbearing potential (WOCBP) must provide a negative urine pregnancy test at screening, and must agree to use a medically accepted and highly effective birth control method (i.e. those with a failure rate less than 1%) for the duration of the study treatment and for 90 days after the final dose of tiragolumab, 5 months after the final dose of atezolizumab, and 6 months after the final dose of cisplatin / 5-fluorouracil (5-FU).

    A woman is considered of childbearing potential ( i.e. fertile) following menarche and until becoming post-menopausal unless permanently sterile. Women will be considered post-menopausal if they have been amenorrhoeic for 12 months without an alternative medical cause. The following age-specific requirements apply:
    1. Amenorrheic for ≥1 year in the absence of chemotherapy and/or hormonal treatments
    2. Luteinizing hormone (LH) and/or follicle stimulating hormone and/or estradiol levels in the post-menopausal range
    3. Radiation induced oophorectomy with last menses >1 year ago
    4. Chemotherapy induced menopause with >1 year interval since last menses
    5. Surgical sterilization (bilateral oophorectomy or hysterectomy)
    6. Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy)
    7. Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
13. For both male and female patients/partners: Contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. Non-sterile males must be willing to use a highly effective method of birth control for the duration of the study treatment and for 90 days after the final dose of tiragolumab, and 6 months after the final dose of cisplatin / 5-FU.

    A sterile male is defined as:
    1. One for whom azoospermia has been previously demonstrated in a semen sample examination as definitive evidence of infertility.
    2. Males with known "low sperm counts" (consistent with "sub-fertility") are not to be considered sterile for purposes of this study.
14. Willingness and ability of patients to comply with the protocol for the duration of the study including undergoing treatment as well as availability for scheduled visits and examinations including follow up.

Exclusion Criteria:

1. Previous or pre-planned potentially curative surgery for the anal carcinoma for the duration of the study. Major surgery (i.e. cystectomy) less than 28 days prior to the first dose of study treatment.
2. Prior treatment for the control of the squamous cell carcinoma of the anal canal. Prior radiotherapy, chemotherapy or treatment with CD137 agonists or immune checkpoint blockade therapies, anti-CTLA-4, anti-TIGIT, anti-PD-1, and anti-PD-L1 therapeutic antibodies are not allowed.
3. History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins. Known hypersensitivity to Chinese hamster ovary cell products or to any component of the tiragolumab or atezolizumab formulation.
4. History of allogeneic stem cell or solid organ transplant.
5. Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis.

   Note: Subjects with the following are not excluded:
   1. Patients with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible for the study.
   2. Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
   3. Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of the following conditions are met:

   i. Rash must cover < 10% of body surface area.

   ii. Disease is well controlled at baseline and requires only low-potency topical corticosteroids.

   iii. There has been no occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months.
6. Subjects that have a diagnosis of immunodeficiency or are receiving systemic steroid therapy or any other form of immunosuppressive therapy within 14 days prior to the first dose of study treatment, with the exceptions:

   1. Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study
   2. Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study.
7. Treatment with investigational therapy within 42 days prior to initiation of study treatment. Observational studies are permitted.
8. Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin 2) within 28 days or 5 drug-elimination half-lives (whichever is longer) prior to first study treatment administration.
9. Not stable treatment with anticoagulant therapies.
10. Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia, or any active infection that could impact patient safety. Active tuberculosis, Epstein-Barr virus(EBV), Hepatitis C virus (HCV), Hepatitis B virus (HBV), or Human immunodeficiency virus (HIV). Current treatment with antiviral therapy for HBV.

    Note: HIV-positive patients may be eligible if they are stable as defined by (a) CD4+ count ≥ 300/μL. (b) Undetectable viral load per standard of care assay. (c) Receiving antiretroviral therapy (ART/HAART) for at least 4 weeks prior to study enrollment, and having not experienced any HIV-related opportunistic infection for at least 4 weeks prior to study enrollment.
11. Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment.

    Note: Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study.
12. Vaccination within 4 weeks of the first dose of study treatment, or anticipation of need for such a vaccine while on trial, and 5 months after last dose of atezolizumab and/or 90 days after last dose of tiragolumab is prohibited except for administration of inactivated vaccines (i.e. SARS-CoV-2 and Influenza vaccines will be permitted).
13. Subject has a history of another uncontrolled malignancy before the first dose of study drug, or any evidence of residual disease from a previously diagnosed malignancy..
14. Presence of the following conditions within the past 6 months:

    1. Uncontrolled diabetes
    2. Uncontrolled or symptomatic hypercalcemia (ionized calcium > 1.5 mmol/L, calcium > 12 mg/dL or corrected serum calcium > ULN)
    3. New York Heart Association class II-IV congestive heart failure
    4. Cerebrovascular accident
    5. Transient ischemic attack
    6. Uncontrolled hypertension
    7. Unstable angina
    8. Myocardial infarction
    9. Grade ≥ 2 peripheral neuropathy as defined by NCI CTCAE v5.0 criteria
    10. Uncontrolled tumor-related pain. Patients requiring pain medication must be on a stable regimen at study entry
    11. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring drainage procedures
15. History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis.
16. Women pregnant or breastfeeding. Fertile and sexually active patients who are not willing to use the appropriate highly effective contraceptive methods.
17. Any underlying medical or psychiatric disorder, which, in the opinion of the investigator, makes the administration of atezolizumab or tiragolumab unsafe or interferes with the informed consent process or trial procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-02-14 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Clinical complete response (CCR) | End of consolidation phase (week 26)
  Clinical complete response (CCR), defined as the percentage of patients who have achieved complete response (CR), disappearance of all lesions according to RECIST 1.1 criteria (locally assessed by the PI) and no presence of residual disease assessed by biopsy at the end of consolidation phase (week 26).
Clinical complete response (CCR) rate | End of consolidation phase (week 26)
  Clinical response rate: Patients will be classified as responders (complete or partial responders) and non-responders based on: 1) the presence of residual disease on tumor biopsy and 2) CT or MRI scans post-treatment (week 26). The binomial proportion and its 95% confidence interval will be used to estimate the CCR rate. Logistic regression analysis will be used to evaluate the effect of baseline characteristics and other covariates with response rate.

SECONDARY OUTCOMES:
Locoregional failure rate (LFR)1 | 1-year after the first dose of study treatment
  locoregional failure rate (LFR), defined as the percentage of patients who present progression/relapse of disease in the anal canal and/or regional organs and/or regional lymph nodes
Locoregional failure rate (LFR)2 | 2 years after the first dose of study treatment
  locoregional failure rate (LFR), defined as the percentage of patients who present progression/relapse of disease in the anal canal and/or regional organs and/or regional lymph nodes
Locoregional failure rate (LFR)3 | 3 years after the first dose of study treatment
  locoregional failure rate (LFR), defined as the percentage of patients who present progression/relapse of disease in the anal canal and/or regional organs and/or regional lymph nodes
Locoregional failure rate (LFR)5 | at the end of study, approximately 5 years after the first dose of study treatment.
  locoregional failure rate (LFR), defined as the percentage of patients who present progression/relapse of disease in the anal canal and/or regional organs and/or regional lymph nodes
Disease-free survival (DFS)1 | 1 year after the first dose of study treatment.
  Disease-free survival (DFS): defined as the time elapsed from the first dose of study treatment to progression, relapse, or death from any cause, whichever occurs first. The investigators will assess the median DFS and the DFS rate at 1, 2, and 3 years, at the end of study (approximately 5 years after the first dose of study treatment). The 1-year, 2-years, and 3-years DFS rates are defined as the rate of patients alive and free of relapse or progression at 1, 2, and 3 years after the first dose of study treatment respectively, estimated by Kaplan-Meier. Patients alive and free of events at the date of the analysis will be censored at their last known tumor assessment.
Disease-free survival (DFS)2 | 2 years after the first dose of study treatment.
  Disease-free survival (DFS): defined as the time elapsed from the first dose of study treatment to progression, relapse, or death from any cause, whichever occurs first. The investigators will assess the median DFS and the DFS rate at 1, 2, and 3 years, at the end of study (approximately 5 years after the first dose of study treatment). The 1-year, 2-years, and 3-years DFS rates are defined as the rate of patients alive and free of relapse or progression at 1, 2, and 3 years after the first dose of study treatment respectively, estimated by Kaplan-Meier. Patients alive and free of events at the date of the analysis will be censored at their last known tumor assessment.
Disease-free survival (DFS)3 | 3 years after the first dose of study treatment.
  Disease-free survival (DFS): defined as the time elapsed from the first dose of study treatment to progression, relapse, or death from any cause, whichever occurs first. The investigators will assess the median DFS and the DFS rate at 1, 2, and 3 years, at the end of study (approximately 5 years after the first dose of study treatment). The 1-year, 2-years, and 3-years DFS rates are defined as the rate of patients alive and free of relapse or progression at 1, 2, and 3 years after the first dose of study treatment respectively, estimated by Kaplan-Meier. Patients alive and free of events at the date of the analysis will be censored at their last known tumor assessment.
Disease-free survival (DFS)5 | And at the end of study, approximately 5 years after the first dose of study treatment.
  Disease-free survival (DFS): defined as the time elapsed from the first dose of study treatment to progression, relapse, or death from any cause, whichever occurs first. The investigators will assess the median DFS and the DFS rate at 1, 2, and 3 years, at the end of study (approximately 5 years after the first dose of study treatment). The 1-year, 2-years, and 3-years DFS rates are defined as the rate of patients alive and free of relapse or progression at 1, 2, and 3 years after the first dose of study treatment respectively, estimated by Kaplan-Meier. Patients alive and free of events at the date of the analysis will be censored at their last known tumor assessment.
Colostomy-free survival (CFS)1 | 1-year after the first dose of study treatment
  Colostomy-free survival (CFS): defined as the time elapsed from the first dose of study treatment to the date the colostomy was required or death from any cause, whichever occurs first. The investigators will assess the median CFS and the CFS rate at 1, 2, and 3 years, and at the end of study (approximately 5 years after the first dose of study treatment). The 1-year, 2-years, and 3-years CFS rates are defined as the rate of patients alive and free of colostomy at 1, 2, and 3 years after the first dose of study treatment respectively, estimated by Kaplan-Meier. Patients alive and free of events at the date of the analysis will be censored at their last known contact.
Colostomy-free survival (CFS)2 | 2-year after the first dose of study treatment
  Colostomy-free survival (CFS): defined as the time elapsed from the first dose of study treatment to the date the colostomy was required or death from any cause, whichever occurs first. The investigators will assess the median CFS and the CFS rate at 1, 2, and 3 years, and at the end of study (approximately 5 years after the first dose of study treatment). The 1-year, 2-years, and 3-years CFS rates are defined as the rate of patients alive and free of colostomy at 1, 2, and 3 years after the first dose of study treatment respectively, estimated by Kaplan-Meier. Patients alive and free of events at the date of the analysis will be censored at their last known contact.
Colostomy-free survival (CFS)3 | 3-year after the first dose of study treatment
  Colostomy-free survival (CFS): defined as the time elapsed from the first dose of study treatment to the date the colostomy was required or death from any cause, whichever occurs first. The investigators will assess the median CFS and the CFS rate at 1, 2, and 3 years, and at the end of study (approximately 5 years after the first dose of study treatment). The 1-year, 2-years, and 3-years CFS rates are defined as the rate of patients alive and free of colostomy at 1, 2, and 3 years after the first dose of study treatment respectively, estimated by Kaplan-Meier. Patients alive and free of events at the date of the analysis will be censored at their last known contact.
Colostomy-free survival (CFS)5 | At the end of study, approximately 5 years after the first dose of study treatment.
  Colostomy-free survival (CFS): defined as the time elapsed from the first dose of study treatment to the date the colostomy was required or death from any cause, whichever occurs first. The investigators will assess the median CFS and the CFS rate at 1, 2, and 3 years, and at the end of study (approximately 5 years after the first dose of study treatment). The 1-year, 2-years, and 3-years CFS rates are defined as the rate of patients alive and free of colostomy at 1, 2, and 3 years after the first dose of study treatment respectively, estimated by Kaplan-Meier. Patients alive and free of events at the date of the analysis will be censored at their last known contact.
Overall survival (OS)3 | 3-years after the first dose of study treatment
  Overall survival (OS): defined as the time elapsed from the first dose of study treatment until death from any cause. The investigators will assess the median OS and the OS rate at 3 and 5 years. The 3-years and 5-years OS rates are defined as the rate of patients alive at 3 and 5 years after the first dose of study treatment respectively, estimated by Kaplan-Meier. Patients alive and free of events at the date of the analysis will be censored at their last known contact.
Overall survival (OS)5 | 5-years after the first dose of study treatment
  Overall survival (OS): defined as the time elapsed from the first dose of study treatment until death from any cause. The investigators will assess the median OS and the OS rate at 3 and 5 years. The 3-years and 5-years OS rates are defined as the rate of patients alive at 3 and 5 years after the first dose of study treatment respectively, estimated by Kaplan-Meier. Patients alive and free of events at the date of the analysis will be censored at their last known contact.
Incidence of adverse events (AEs) | Throughout the study period, approximately 5 years per patient
  To evaluate safety of the intended treatment regimen based on the frequency and severity of adverse events (AE) assessed by NCI CTCAE v5.0. Incidence of adverse events (AEs) evaluated as percentage of patients experiencing an adverse event.
Incidence of Treatment-emergent adverse events (TEAEs) | Throughout the study period, approximately 5 years per patient
  To evaluate safety of the intended treatment regimen based on the frequency and severity of Treatment-emergent adverse events (TEAEs) assessed by NCI CTCAE v5.0. Incidence of Treatment-emergent adverse events (TEAEs) evaluated as percentage of patients experiencing an treatment-emergent adverse events.

OTHER OUTCOMES:
Health-related quality of life (HRQoL) | concomitant phase (week1); consolidation phase (week 7) and after the end of treatment (week 24)
  The EORTC QLQ-C30 questionnaire is a specific questionnaire validated for cancer that is composed of 30 questions or items. The questionnaire is structured in 5 functional scales (physical functioning, daily activities, emotional functioning, cognitive functioning and social functioning), 3 symptom scales (fatigue, pain and nausea, vomiting), 1 global health status scale, and 6 independent items (dyspnea, insomnia, anorexia, constipation, diarrhea and economic impact). Values between 1 and 4 (1: not at all, 2: a little, 3: quite, 4: a lot) are assigned according to the patient's responses to the item, only in items 29 and 30 are they evaluated with a score of 1 to 7 (1: dreadful, 7: excellent). The scores obtained are standardized and a score between 0 and 100 is obtained, which determines the level of impact of the cancer on the patient on each of the scales. A higher score indicating a better HRQoL.
Determination of the most frequent molecular alterations in this pathology | During the screening, and after the end of treatment (Week 26).
  Percentage of patients presenting alterations or deregulation in any of the following (composite endpoint)
  * The expression of immune checkpoint proteins (PD-1, PD-L1, CD28, OX40, CD40, or others) in blood and tumor samples.
  * The expression of potential molecular biomarkers (HPV, KRAS, TP53) in liquid biopsy (ctDNA) and tumor samples.
  * The expression of poliovirus receptor (PVR) and HPV status.
  * The presence of infiltrating T cell lymphocytes (CD45, CD3, CD8, CD4, CD56, IFNbeta, STAT1,CD 163, H2AX, or others) in tumor samples.
  * The T-cell clonality (TCR) in blood samples
  * The presence of ctDNA in blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Jaume Capdevila, Study Chair — Hospital Vall d'Hebron
Locations (15):
- Spain (15):
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Institut Català d'Oncologia (ICO) Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital Arnau de Vilanova, Lleida, Barcelona
  - Hospital Sant Joan Despí, Martorell, Barcelona
  - Consorcio Corporación Sanitaria Parc Taulí, Sabadell, Barcelona
  - Hospital General Universitario de Toledo, Toledo, Castille-La Mancha
  - HU Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital General de Ciudad Real, Ciudad Real
  - Complejo Asistencial Universitario de León, León
  - Hospital Universitario 12 de Octubre, Madrid
  - Consorcio Hospital General Universitario de Valencia, Valencia
  - Hospital Universitario y Politécnico la Fe de Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) anonymized could be shared upon request if the use is within the scope and protection level authorized by the patients by the signature of the informed consent